CLINICAL TRIAL: NCT04995029
Title: A Randomised, Double-Blind Study Comparing 2 Maintenance Dosing Regimens of Buprenorphine Extended-Release Subcutaneous Injection (RBP-6000) in Treatment-Seeking Adult Participants With Opioid Use Disorder and High-risk Opioid Use
Brief Title: Buprenorphine Extended-Release Subcutaneous Injection (RBP-6000) in High-risk Users
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INDV-6000-401; TRANSFORM (Other: Indivior)
Record Dates: First submitted 2021-07-29; First posted 2021-08-06 (Actual); Results first posted 2025-09-25 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Moderate to Severe Opioid-use Disorder
MeSH Terms: interventions — Sublocade

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The induction phase of the study will be open label. The maintenance phase of the study will be conducted in a double-blind manner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Induction Phase: Rapid Induction (Experimental): Participants will receive 4 mg transmucosal buprenorphine on Day 1. Participants meeting eligibility requirements will then receive 300 mg extended-release buprenorphine by subcutaneous injection at least 1 hour later and a second dose on Day 8.
  Interventions: Drug: Transmucosal Buprenorphine; Drug: Extended-release Buprenorphine
- Induction Phase: Standard of Care Induction (Experimental): Participants will receive transmucosal buprenorphine for a minimum of 7 days per applicable product labelling information. Participants meeting eligibility requirements will receive 300 mg extended-release buprenorphine by subcutaneous injection on Day 1 and a second dose on Day 8.
  Interventions: Drug: Transmucosal Buprenorphine; Drug: Extended-release Buprenorphine
- Maintenance Phase: Extended-release Buprenorphine 100 mg (Experimental): Participants eligible to continue treatment will be randomized at Week 6 to receive maintenance doses of 100 mg extended-release buprenorphine by subcutaneous injection every 4 weeks for a total of up to 8 maintenance injections (Weeks 6 to 34).
  Interventions: Drug: Extended-release Buprenorphine
- Maintenance Phase: Extended-release Buprenorphine 300 mg (Experimental): Participants eligible to continue treatment will be randomized at Week 6 to receive maintenance doses of 300 mg extended-release buprenorphine by subcutaneous injection every 4 weeks for a total of up to 8 maintenance injections (Weeks 6 to 34).
  Interventions: Drug: Extended-release Buprenorphine

INTERVENTIONS:
Drug: Transmucosal Buprenorphine — Transmucosal (TM) buprenorphine as selected by the Investigator per local prescribing guidelines, administered either under the tongue (sublingual) or between the gum and cheek (buccal)
  Arms: Induction Phase: Rapid Induction; Induction Phase: Standard of Care Induction
Drug: Extended-release Buprenorphine — Administered by subcutaneous injection
  Other Names: RBP-6000; SUBLOCADE

SUMMARY:
The primary objective of the induction phase of the study is to compare treatment retention of participants following rapid induction or standard of care (SoC) induction onto extended-release buprenorphine.

The primary objective of the maintenance phase is to compare the efficacy of 100 mg and 300 mg maintenance doses of extended-release buprenorphine administered every 4 weeks.

DETAILED DESCRIPTION:
This study consists of an open-label induction phase followed by a double-blind maintenance phase. Each phase is designed to test separate objectives and endpoints.

In the induction phase participants who use opioids via an injection route and/or use high doses of opioids who are in withdrawal will be randomly assigned in a 2:1 ratio to extended-release buprenorphine rapid induction or SoC induction. The rapid induction arm is designed to initiate extended-release buprenorphine treatment following a single dose of transmucosal (TM) buprenorphine, while the SoC induction arm inducts the participant onto extended-release buprenorphine using a TM buprenorphine-containing product for a minimum of 7 days. All participants will receive the first injection of extended-release buprenorphine on Day 1 and the second injection on Day 8.

Participants eligible to continue treatment in the maintenance phase will be randomized at Week 6 prior to Injection 3 in a 1:1 ratio to receive maintenance doses of either 300 mg or 100 mg extended-release buprenorphine every 4 weeks for a total of up to 8 maintenance injections.

ELIGIBILITY:
Inclusion Criteria:

1. Has signed the informed consent form (ICF) and is able and willing to comply with the requirements and restrictions listed therein.
2. Is 18 years of age or older at the time of signing the ICF.
3. Currently meets Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria for moderate or severe opioid use disorder (OUD).
4. Has a history of OUD as defined by documented medical history of OUD for at least 90 days immediately prior to providing informed consent.
5. Meets at least 1 of these criteria for high-risk opioid use at the Screening visit:

   1. using opioids via the injection route for an average of 5 or more days per week in the last 4 weeks.
   2. using at least 500 mg IV heroin equivalent (e.g., 1250 mg intravenous (IV) morphine) or self-reported use of any dose of highly potent synthetic opioids (fentanyl and analogues excluding transdermal patches) for an average of 5 or more days per week in the last 4 weeks by any route.
6. Is seeking medication for the treatment of OUD.
7. Is an appropriate candidate for opioid partial-agonist medications for opioid use disorder (MOUD) in the opinion of the Investigator or medically qualified sub-Investigator.
8. Agrees not to use buprenorphine-containing products other than those administered as part of study treatment for the duration of the treatment period.
9. A female participant is eligible to participate if she is not pregnant, not lactating and, if of childbearing potential, agrees not to become pregnant while on the study and to use medically acceptable means of contraception while on the study).

Exclusion Criteria:

1. Has current diagnosis, other than OUD, requiring chronic opioid treatment.
2. Has concurrent primary substance use disorder, as defined by DSM-5 criteria, other than opioid, tobacco, cannabis or alcohol use disorders.
3. Meets DSM-5 criteria for severe alcohol use disorder.
4. Has had significant traumatic injury or major surgical procedure (as defined by the Investigator) within 30 days prior to the first dose of RBP-6000 or still recovering from prior such injury or surgery.
5. Has congenital long QT syndrome, history of prolonged QT in the 3 months prior to Screening, or history of medications or other factors that are at risk for Torsades de Pointes.
6. Has abdominal area unsuitable for subcutaneous injections (e.g., nodules, scarring, lesions, excessive pigment).
7. Has history of suicidal ideation within 30 days prior to informed consent or history of a suicide attempt in the 6 months prior to informed consent.
8. Has uncontrolled intercurrent illness including, but not limited to, a medical or psychiatric illness/social situation that would limit compliance with study requirements or compromise the ability of the participant to provide written informed consent.
9. Has any other active medical condition, organ disease or concurrent medication or treatment that may either compromise participant safety or interfere with study endpoints.
10. Has total bilirubin ≥ 1.5 × upper limit of normal (ULN) (with direct bilirubin > 1.3 mg/dL), alanine aminotransferase (ALT) ≥ 3 × ULN, aspartate aminotransferase (AST) ≥ 3 × ULN, serum creatinine > 2 × ULN, or international normalized ratio (INR) > 1.5 × ULN at Screening.
11. Has known allergy or hypersensitivity to buprenorphine or any component of the ATRIGEL Delivery System.
12. Is undergoing concurrent or has had prior treatment with any long-acting form of buprenorphine-containing product in the past 2 years, or if > 2 years has a positive UDS for buprenorphine at screening; treatment with oral buprenorphine, oral naltrexone or methadone products within 14 days prior to consent; or treatment with depot naltrexone within the 3 months prior to consent.
13. Is undergoing concurrent treatment with another investigational agent or enrollment in another clinical study (except for an observational study) or treatment with another investigational agent within 30 days prior to Screening.
14. Is undergoing concurrent treatment with medications contraindicated for use with buprenorphine as per local prescribing information.
15. Has any pending legal status or pending legal action that could prohibit full participation in or compliance with study procedures.
16. Is under court order requiring treatment for OUD.
17. Is a member of site staff and/or has a financial interest in Indivior, or is an immediate family member of either the site staff and/or Indivior employee, directly involved in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 785 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Director Clinical Development, Study Director — Indivior Inc.
Locations (29):
- United States (28):
  - Collaborative Neuroscience Network, LLC, Garden Grove, California
  - Asclepes Research Centers, Panorama City, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Bay Pines VA Healthcare System, Bay Pines, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Accel Research Sites- Lakeland Clinical Research Unit, Lakeland, Florida
  - Behavioral Clinical Research, Inc, Miami Lakes, Florida
  - Innovative Clinical Research Inc., North Miami, Florida
  - Clinical Neuroscience Solutions, Inc, Orlando, Florida
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Hassman Research Institute, Berlin, New Jersey
  - Center For Emotional Fitness, Cherry Hill, New Jersey
  - ICAHN School of Medicine at Mount Sinai, New York, New York
  - Duke Hospital, Durham, North Carolina
  - Monroe Biomedical Research, Monroe, North Carolina
  - Midwest Clinical Research, Dayton, Ohio
  - Pahl Pharmaceutical Professionals LLC, Oklahoma City, Oklahoma
  - SP Research, PLLC, Oklahoma City, Oklahoma
  - Unity Clinical Research, Oklahoma City, Oklahoma
  - Today Clinical Research, Oklahoma City, Oklahoma
  - Clinical Research Associates of Central PA, Altoona, Pennsylvania
  - Carolina Medical Research, LLC, Clinton, South Carolina
  - Prisma Health ITOR Research Pharmacy, Greenville, South Carolina
  - Carolina Medical Research, LLC, Greenville, South Carolina
  - David Weitzman, Myrtle Beach, South Carolina
  - Insite Clinical Research, DeSoto, Texas
  - Progressive Clinical Research, Bountiful, Utah
  - Alpine Research Organization, Clinton, Utah
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lan Q, He X, Costa D, Tian W. [Glutathione S-transferase GSTM1 and GSTT1 genotypes and susceptibility to lung cancer]. Wei Sheng Yan Jiu. 1999 Jan 30;28(1):9-11. Chinese. PMID 12712736
- [Result] Shiwach R, Le Foll B, Alho H, Dunn KE, Strafford S, Zhao Y, Dobbins RL. Rapid vs Standard Induction to Injectable Extended-Release Buprenorphine: A Randomized Clinical Trial. JAMA Netw Open. 2025 Oct 1;8(10):e2537319. doi: 10.1001/jamanetworkopen.2025.37319. PMID 41085986
- [Derived] Shiwach R, Le Foll B, Alho H, Dunn KE, Strafford S, Zhao Y, Dobbins RL. Comparison of Extended-Release Buprenorphine Doses for Treating High-Risk Opioid Use: A Randomized Clinical Trial. JAMA Netw Open. 2025 Dec 1;8(12):e2548043. doi: 10.1001/jamanetworkopen.2025.48043. PMID 41405885

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Period was 26 Oct 2021 to 26 Jun 2024.
Pre-assignment Details: Induction Phase: Participants were required to be in withdrawal (COWS score ≥8) to receive transmucosal (TM) buprenorphine (BUP).
  To receive RBP-6000, the participant did not display any allergic/ hypersensitivity reaction to TM BUP, did not experience precipitated withdrawal symptoms from the most recent TM BUP administration that would prevent RBP-6000 injection, and was not sedated.
  For standard of care, the participant had been dose-adjusted onto TM BUP for ≥7 days.
Groups:
- Induction Phase: Rapid Induction: Participants will receive 4 mg transmucosal buprenorphine on Day 1. Participants meeting eligibility requirements will then receive 300 mg extended-release buprenorphine by subcutaneous injection at least 1 hour later and a second dose on Day 8.
  Participants are followed until Injection 3 (Week 6).
  Transmucosal Buprenorphine: Transmucosal (TM) buprenorphine as selected by the Investigator per local prescribing guidelines, administered either under the tongue (sublingual) or between the gum and cheek (buccal)
  Extended-release Buprenorphine: Administered by subcutaneous injection
- Induction Phase: Standard of Care Induction: Participants will receive transmucosal buprenorphine for a minimum of 7 days per applicable product labelling information. Participants meeting eligibility requirements will receive 300 mg extended-release buprenorphine by subcutaneous injection on Day 1 and a second dose on Day 8.
  Participants are followed until Injection 3 (Week 6).
  Transmucosal Buprenorphine: Transmucosal (TM) buprenorphine as selected by the Investigator per local prescribing guidelines, administered either under the tongue (sublingual) or between the gum and cheek (buccal)
  Extended-release Buprenorphine: Administered by subcutaneous injection
- Maintenance Phase: Extended-release Buprenorphine 100 mg: Participants eligible to continue treatment will be randomized at Week 6 to receive maintenance doses of 100 mg extended-release buprenorphine by subcutaneous injection every 4 weeks for a total of up to 8 maintenance injections (Weeks 6 to 34).
  Participants are followed until Week 38.
  Extended-release Buprenorphine: Administered by subcutaneous injection
- Maintenance Phase: Extended-release Buprenorphine 300 mg: Participants eligible to continue treatment will be randomized at Week 6 to receive maintenance doses of 300 mg extended-release buprenorphine by subcutaneous injection every 4 weeks for a total of up to 8 maintenance injections (Weeks 6 to 34).
  Participants are followed until Week 38.
  Extended-release Buprenorphine: Administered by subcutaneous injection
Period: Induction Phase
Arm/Group | Induction Phase: Rapid Induction | Induction Phase: Standard of Care Induction | Maintenance Phase: Extended-release Buprenorphine 100 mg | Maintenance Phase: Extended-release Buprenorphine 300 mg
Started (Open-label Randomized) | 518 | 267 | 0 | 0
Received TM BUP | 513 | 264 | 0 | 0
Received RBP-6000 Injection 1 | 444 | 159 | 0 | 0
Received RBP-6000 Injection 2 | 339 | 145 | 0 | 0
Completed (Completed/Received RBP-6000 Injection 3) | 298 | 137 | 0 | 0
Not Completed | 220 | 130 | 0 | 0
Not completed — Did not meet eligibility criteria | 5 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 85 | 42 | 0 | 0
Not completed — Lost to Follow-up | 103 | 67 | 0 | 0
Not completed — Adverse Event | 5 | 3 | 0 | 0
Not completed — Physician Decision | 11 | 8 | 0 | 0
Not completed — Incarceration | 6 | 3 | 0 | 0
Not completed — Not otherwise described | 5 | 5 | 0 | 0
Period: Maintenance Phase
Arm/Group | Induction Phase: Rapid Induction | Induction Phase: Standard of Care Induction | Maintenance Phase: Extended-release Buprenorphine 100 mg | Maintenance Phase: Extended-release Buprenorphine 300 mg
Started (Treated with maintenance dose in Double-blind Treatment Period) | 0 | 0 | 218 | 217
Completed (Completed DBTP End of Treatment Week 38) | 0 | 0 | 134 | 128
Not Completed | 0 | 0 | 84 | 89
Not completed — Lost to Follow-up | 0 | 0 | 51 | 44
Not completed — Did not meet eligibility criteria | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 8 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 17 | 31
Not completed — Incarceration | 0 | 0 | 4 | 3
Not completed — Not otherwise described | 0 | 0 | 2 | 3
Not completed — Pregnancy | 0 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: In the Induction Phase, of the 785 participants randomized (Substudy Randomized Population [SRP]), 729 were included in the Substudy Full Analysis Set (SFAS), the analysis set used for most endpoints and all safety analyses. Compared with the SRP, the SFAS excluded 56 participants: 48 who were randomized and inducted with neither rapid induction nor standard of care injection (which was a key protocol deviation) as well as 8 participants who discontinued prior to receiving TM buprenorphine.
Groups:
- Total: Total of all reporting groups
Arm/Group | Induction Phase: Rapid Induction | Induction Phase: Standard of Care Induction | Maintenance Phase: Extended-release Buprenorphine 100 mg | Maintenance Phase: Extended-release Buprenorphine 300 mg | Total
Number analyzed (Participants) | 474 | 255 | 218 | 217 | 1164
Age, Categorical [Count of Participants; unit: Participants] — Population: The number analyzed differs from overall because baseline data are presented separately for the Induction Phase and the Maintenance Phase.
  Participants
    Induction Phase: number analyzed (Participants) | 474 | 255 | 0 | 0 | 729
    Induction Phase: <=18 years | 1 | 1 | 0 | 0 | 2
    Induction Phase: Between 18 and 65 years | 470 | 252 | 0 | 0 | 722
    Induction Phase: >=65 years | 3 | 2 | 0 | 0 | 5
    Maintenance Phase: number analyzed (Participants) | 0 | 0 | 218 | 217 | 435
    Maintenance Phase: <=18 years | 0 | 0 | 0 | 0 | 0
    Maintenance Phase: Between 18 and 65 years | 0 | 0 | 216 | 214 | 430
    Maintenance Phase: >=65 years | 0 | 0 | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The number analyzed differs from overall because baseline data are presented separately for the Induction Phase and the Maintenance Phase.
  years
    Induction Phase: number analyzed (Participants) | 474 | 255 | 0 | 0 | 729
    Induction Phase | 40.9 (10.68) | 40.4 (9.77) |  |  | 40.7 (10.37)
    Maintenance Phase: number analyzed (Participants) | 0 | 0 | 218 | 217 | 435
    Maintenance Phase |  |  | 41.5 (10.58) | 41.7 (11.17) | 41.6 (10.87)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The number analyzed differs from overall because baseline data are presented separately for the Induction Phase and the Maintenance Phase.
  Participants
    Induction Phase: number analyzed (Participants) | 474 | 255 | 0 | 0 | 729
    Induction Phase: Female | 202 | 121 | 0 | 0 | 323
    Induction Phase: Male | 272 | 134 | 0 | 0 | 406
    Maintenance Phase: number analyzed (Participants) | 0 | 0 | 218 | 217 | 435
    Maintenance Phase: Female | 0 | 0 | 95 | 92 | 187
    Maintenance Phase: Male | 0 | 0 | 123 | 125 | 248
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The number analyzed differs from overall because baseline data are presented separately for the Induction Phase and the Maintenance Phase.
  Participants
    Induction Phase: number analyzed (Participants) | 474 | 255 | 0 | 0 | 729
    Induction Phase: Hispanic or Latino | 76 | 32 | 0 | 0 | 108
    Induction Phase: Not Hispanic or Latino | 394 | 220 | 0 | 0 | 614
    Induction Phase: Unknown or Not Reported | 4 | 3 | 0 | 0 | 7
    Maintenance Phase: number analyzed (Participants) | 0 | 0 | 218 | 217 | 435
    Maintenance Phase: Hispanic or Latino | 0 | 0 | 25 | 37 | 62
    Maintenance Phase: Not Hispanic or Latino | 0 | 0 | 191 | 178 | 369
    Maintenance Phase: Unknown or Not Reported | 0 | 0 | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The number analyzed differs from overall because baseline data are presented separately for the Induction Phase and the Maintenance Phase.
  Participants
    Induction Phase: number analyzed (Participants) | 474 | 255 | 0 | 0 | 729
    Induction Phase: American Indian or Alaska Native | 4 | 2 | 0 | 0 | 6
    Induction Phase: Asian | 1 | 0 | 0 | 0 | 1
    Induction Phase: Native Hawaiian or Other Pacific Islander | 4 | 1 | 0 | 0 | 5
    Induction Phase: Black or African American | 85 | 37 | 0 | 0 | 122
    Induction Phase: White | 358 | 207 | 0 | 0 | 565
    Induction Phase: More than one race | 0 | 0 | 0 | 0 | 0
    Induction Phase: Unknown or Not Reported | 22 | 8 | 0 | 0 | 30
    Maintenance Phase: number analyzed (Participants) | 0 | 0 | 218 | 217 | 435
    Maintenance Phase: American Indian or Alaska Native | 0 | 0 | 5 | 1 | 6
    Maintenance Phase: Asian | 0 | 0 | 0 | 1 | 1
    Maintenance Phase: Native Hawaiian or Other Pacific Islander | 0 | 0 | 2 | 1 | 3
    Maintenance Phase: Black or African American | 0 | 0 | 46 | 48 | 94
    Maintenance Phase: White | 0 | 0 | 160 | 154 | 314
    Maintenance Phase: More than one race | 0 | 0 | 0 | 0 | 0
    Maintenance Phase: Unknown or Not Reported | 0 | 0 | 5 | 12 | 17
Body Mass Index (kg/m2) [Mean (Standard Deviation); unit: kg/m2] — Population: The number analyzed differs from overall because baseline data are presented separately for the Induction Phase and the Maintenance Phase.
  kg/m2
    Induction Phase: number analyzed (Participants) | 474 | 255 | 0 | 0 | 729
    Induction Phase | 26.83 (5.969) | 27.05 (6.305) |  |  | 26.91 (6.085)
    Maintenance Phase: number analyzed (Participants) | 0 | 0 | 218 | 217 | 435
    Maintenance Phase |  |  | 26.96 (6.446) | 26.53 (5.860) | 26.75 (6.157)
Opioids Lifetime Use (years) [Mean (Standard Deviation); unit: years] — Population: The number analyzed differs from overall because baseline data are presented separately for the Induction Phase and the Maintenance Phase.
  years
    Induction Phase: number analyzed (Participants) | 474 | 255 | 0 | 0 | 729
    Induction Phase | 14.8 (9.77) | 14.6 (9.37) |  |  | 14.7 (9.62)
    Maintenance Phase: number analyzed (Participants) | 0 | 0 | 218 | 217 | 435
    Maintenance Phase |  |  | 14.8 (9.80) | 15.8 (10.84) | 15.3 (10.33)
Opioid Use Last 4 Weeks (days) [Mean (Standard Deviation); unit: days] — Population: The number analyzed differs from overall because baseline data are presented separately for the Induction Phase and the Maintenance Phase.
  days
    Induction Phase: number analyzed (Participants) | 474 | 255 | 0 | 0 | 729
    Induction Phase | 27.8 (1.10) | 27.7 (1.28) |  |  | 27.8 (1.17)
    Maintenance Phase: number analyzed (Participants) | 0 | 0 | 218 | 217 | 435
    Maintenance Phase |  |  | 27.7 (1.36) | 27.8 (0.89) | 27.8 (1.15)
Previous Opioid Overdose (Yes) [Count of Participants; unit: Participants] — Population: The number analyzed differs from overall because baseline data are presented separately for the Induction Phase and the Maintenance Phase.
  Participants
    Induction Phase: number analyzed (Participants) | 474 | 255 | 0 | 0 | 729
    Induction Phase | 158 | 85 | 0 | 0 | 243
    Maintenance Phase: number analyzed (Participants) | 0 | 0 | 218 | 217 | 435
    Maintenance Phase | 0 | 0 | 69 | 74 | 143
Fentanyl UDS Result at Induction Day 1 Visit [Count of Participants; unit: Participants] — Population: The number analyzed differs from overall because baseline data are presented separately for the Induction Phase and the Maintenance Phase.
  Participants
    Induction Phase: number analyzed (Participants) | 474 | 255 | 0 | 0 | 729
    Induction Phase | 367 | 196 | 0 | 0 | 563
    Maintenance Phase: number analyzed (Participants) | 0 | 0 | 218 | 217 | 435
    Maintenance Phase | 0 | 0 | 153 | 170 | 323
Detoxed From Opioids Previously (Yes) [Count of Participants; unit: Participants] — Population: The number analyzed differs from overall because baseline data are presented separately for the Induction Phase and the Maintenance Phase.
  Participants
    Induction Phase: number analyzed (Participants) | 474 | 255 | 0 | 0 | 729
    Induction Phase | 354 | 193 | 0 | 0 | 547
    Maintenance Phase: number analyzed (Participants) | 0 | 0 | 218 | 217 | 435
    Maintenance Phase | 0 | 0 | 159 | 165 | 324
Using Opioids Via Injection Route for Average of ≥5 Days Per Week in the Last 4 Weeks [Count of Participants; unit: Participants] — Population: The number analyzed differs from overall because baseline data are presented separately for the Induction Phase and the Maintenance Phase.
  Participants
    Induction Phase: number analyzed (Participants) | 474 | 255 | 0 | 0 | 729
    Induction Phase | 136 | 78 | 0 | 0 | 214
    Maintenance Phase: number analyzed (Participants) | 0 | 0 | 218 | 217 | 435
    Maintenance Phase | 0 | 0 | 80 | 77 | 157
Main Route of Opioid Use Last 4 Weeks [Count of Participants; unit: Participants] — Population: The number analyzed differs from overall because baseline data are presented separately for the Induction Phase and the Maintenance Phase.
  Participants
    Induction Phase: number analyzed (Participants) | 474 | 255 | 0 | 0 | 729
    Induction Phase: Injection | 131 | 79 |  |  | 210
    Induction Phase: Smoking | 218 | 109 |  |  | 327
    Induction Phase: Oral | 9 | 6 |  |  | 15
    Induction Phase: Snorting | 114 | 60 |  |  | 174
    Induction Phase: Other | 2 | 1 |  |  | 3
    Maintenance Phase: number analyzed (Participants) | 0 | 0 | 218 | 217 | 435
    Maintenance Phase: Injection |  |  | 62 | 59 | 121
    Maintenance Phase: Smoking |  |  | 92 | 94 | 186
    Maintenance Phase: Oral |  |  | 2 | 8 | 10
    Maintenance Phase: Snorting |  |  | 62 | 55 | 117
    Maintenance Phase: Other |  |  | 0 | 1 | 1
Multiple Drug Class Use - Last 4 Weeks at Screening Self-report or UDS Prior to First DB Injection [Count of Participants; unit: Participants] — Multiple Drug Class Use - Last 4 Weeks at Screening Self-report or UDS Prior to First DB Injection data were analyzed only for the main study (ie, reflected in the Maintenance Phase arms). Population: The number analyzed differs from overall because baseline data are presented separately for the Induction Phase and the Maintenance Phase.
  Participants
    number analyzed (Participants) | 0 | 0 | 218 | 217 | 435
    (all) |  |  | 217 | 213 | 430
Fentanyl + Any Other Drug Class on Screening UDS [Count of Participants; unit: Participants] — Fentanyl + Any Other Drug Class on Screening UDS data were analyzed only for the main study (ie, reflected in the Maintenance Phase arms). Population: The number analyzed differs from overall because baseline data are presented separately for the Induction Phase and the Maintenance Phase.
  Participants
    number analyzed (Participants) | 0 | 0 | 218 | 217 | 435
    (all) |  |  | 142 | 151 | 293
Used Fentanyl ≥14 Times/Week in the Last 7 Days Prior to Screening [Count of Participants; unit: Participants] — High-frequency fentanyl use was analyzed only for the main study (ie, reflected in the Maintenance Phase arms). Population: The number analyzed differs from overall because baseline data are presented separately for the Induction Phase and the Maintenance Phase.
  Participants
    number analyzed (Participants) | 0 | 0 | 218 | 217 | 435
    (all) |  |  | 88 | 104 | 192
Used Fentanyl Daily in the Last 7 Days at Screening [Count of Participants; unit: Participants] — High-frequency fentanyl use was analyzed only for the main study (ie, reflected in the Maintenance Phase arms). Population: The number analyzed differs from overall because baseline data are presented separately for the Induction Phase and the Maintenance Phase.
  Participants
    number analyzed (Participants) | 0 | 0 | 218 | 217 | 435
    (all) |  |  | 98 | 111 | 209
Used Fentanyl ≥14 Times/Week AND Daily in the Last 7 Days Prior to Screening [Count of Participants; unit: Participants] — High-frequency fentanyl use was analyzed only for the main study (ie, reflected in the Maintenance Phase arms). Population: The number analyzed differs from overall because baseline data are presented separately for the Induction Phase and the Maintenance Phase.
  Participants
    number analyzed (Participants) | 0 | 0 | 218 | 217 | 435
    (all) |  |  | 73 | 90 | 163

OUTCOME MEASURES:

1. Primary Outcome: Maintenance Phase: Percentage of Responders for Weekly Opioid Use Over Weeks 20 to 38
Description: A responder for weekly opioid use is defined as a participant whose percentage of visits with opioid abstinence is greater than or equal to 80% over Weeks 20 to 38 inclusive.
  Opioid abstinence is defined as a negative urine drug screen (UDS) result and negative responses to the TimeLine Follow Back (TLFB) interview for opioid use. The TLFB asks participants to retrospectively estimate their daily drug use for each of the past 7 days prior to the visit.
Time Frame: Weeks 20 to 38
Population: The Full Analysis Set (FAS): Participants who met all inclusion/exclusion criteria, were randomized, and received at least 1 maintenance RBP-6000 injection post DB Randomization. Participants were analyzed according to the randomized treatment arm. This population served as the primary analysis population for efficacy analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Phase: Extended-release Buprenorphine 100 mg | Maintenance Phase: Extended-release Buprenorphine 300 mg
Number analyzed (Participants) | 218 | 216
Participants | 44 | 50
Statistical Analysis 1: Comparison: Maintenance Phase: Extended-release Buprenorphine 100 mg vs Maintenance Phase: Extended-release Buprenorphine 300 mg; Based on Phase 3 results, for the primary efficacy endpoint of INDV-6000-401, a sample size of 195 per arm was estimated to provide approximately 90% power at 2-sided 0.05 alpha level to detect a difference of 15.6%. Since the participant population in this study had more severe OUD compared with the Phase 3 DB study, the responder rates and treatment differences were anticipated to be lower; Test type: Superiority — Any missed or skipped visit was counted as non-negative or de-facto positive. Difference between DB treatment arms was compared using CMH test accounting for randomization stratification (Opioid injection: Yes/No, Week 6 UDS Fentanyl result: Positive/Negative). Statistical superiority was declared if CMH weighted difference in proportion of responders in the 300-mg arm minus the proportion of responders in the 100-mg arm was >0 and the 2-sided P-value of CMH test ≤0.05; p = 0.4819, Cochran-Mantel-Haenszel — CMH weighted treatment difference and P-value based on CMH randomization stratified analysis using Sato (1989) variance equation. Treatment difference estimate calculated as weighted average of strata-specific estimates within each analysis stratum; Difference between DB treatment arms was compared using CMH test accounting for randomization stratification; CMH treatment difference = 2.62, 95% CI 2-sided [-4.69 to 9.93]
Statistical Analysis 2: Comparison: Maintenance Phase: Extended-release Buprenorphine 100 mg vs Maintenance Phase: Extended-release Buprenorphine 300 mg; Post-hoc subgroup analyses of the primary endpoint to characterize the population of patients who would benefit from the higher maintenance dosing regimen identified participants who reported using fentanyl ≥14 times per week at Screening as one such group; Test type: Superiority — [test comment as in outcome 1, analysis 1]; CMH treatment difference = 12.24, 95% CI 2-sided [2.35 to 22.12] — CMH weighted treatment difference based on CMH randomization stratified analysis using Sato (1989) variance equation. Treatment difference estimate calculated as weighted average of strata-specific estimates within each analysis stratum; The posterior possibility of responder rate difference (300 mg-100 mg) >0 was estimated (via Bayesian beta-binomial model using non-informative uniform prior, ie, Beta (1,1), within individual treatment groups) to evaluate the superiority of 300 mg over 100 mg. Bayesian posterior probability of superiority 300-mg dose to 100-mg dose=99.099%
Statistical Analysis 3: Comparison: Maintenance Phase: Extended-release Buprenorphine 100 mg vs Maintenance Phase: Extended-release Buprenorphine 300 mg; Post-hoc subgroup analyses of the primary endpoint to characterize the population of patients who would benefit from the higher maintenance dosing regimen identified participants who reported using fentanyl daily at Screening as one such group; Test type: Superiority — [test comment as in outcome 1, analysis 1]; CMH treatment difference = 11.06, 95% CI 2-sided [0.36 to 21.56] — CMH weighted treatment difference and P-value based on CMH randomization stratified analysis using Sato (1989) variance equation. Treatment difference estimate calculated as weighted average of strata-specific estimates within each analysis stratum; The posterior possibility of responder rate difference (300 mg-100 mg) >0 was estimated (via Bayesian beta-binomial model using non-informative uniform prior, ie, Beta (1,1), within individual treatment groups) to evaluate the superiority of 300 mg over 100 mg. Bayesian posterior probability of superiority of 300-mg dose to 100-mg dose=97.846%
Statistical Analysis 4: Comparison: Maintenance Phase: Extended-release Buprenorphine 100 mg vs Maintenance Phase: Extended-release Buprenorphine 300 mg; Post-hoc subgroup analyses of the primary endpoint to characterize the population of patients who would benefit from the higher maintenance dosing regimen identified participants who reported using fentanyl ≥14 times per week AND daily at Screening as one such group; Test type: Superiority — [test comment as in outcome 1, analysis 1]; CMH treatment difference = 15.37, 95% CI 2-sided [4.61 to 26.09] — [estimate comment as in outcome 1, analysis 2]; The posterior possibility of responder rate difference (300 mg-100 mg) >0 was estimated (via Bayesian beta-binomial model using non-informative uniform prior, ie, Beta (1,1), within individual treatment groups) to evaluate the superiority of 300 mg over 100 mg. Bayesian posterior probability of superiority of 300-mg dose to 100-mg dose=99.675%

2. Primary Outcome: Induction Phase: Percentage of Participants Receiving Injection 2 at the Week 2 Visit
Description: Treatment retention at Injection 2 was defined as the proportion of participants receiving Injection 2 at the Week 2 Visit among those in the Evaluable Population for Treatment Retention/Discontinuation. Participants who received Injection 2 at Week 2 (nominal) Visit and those who missed Injection 2 at Week 2 (nominal) Visit but received Injection 3 at the Week 6 Day 36 Visit were counted as "Yes" for treatment retention at Injection 2; otherwise, participants were counted as "No".
Time Frame: Week 2
Population: Evaluable Population for Treatment Retention/Discontinuation: For analysis pertaining to treatment retention and time to treatment discontinuation, the Substudy Full Analysis Set participants who discontinued treatment due to not meeting inclusion/exclusion criteria were also excluded. The participants were analyzed corresponding to the induction arm they received ("as treated", ie, actual arm).
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Phase: Rapid Induction | Induction Phase: Standard of Care Induction
Number analyzed (Participants) | 470 | 253
Participants | 312 | 138
Statistical Analysis 1: Comparison: Induction Phase: Rapid Induction vs Induction Phase: Standard of Care Induction; Null and alternative statistical hypotheses: H0: retention rate of RI - SoC induction≤-10% (non-inferiority [NI] margin of 10%) HA: retention rate of RI-SoC induction>-10%. Criterion for success (ie, demonstrating non-inferiority [NI]) was based on posterior probability of retention rate difference (RI-SoC)>-10%. NI of RI to SoC induction was declared if the posterior probability was higher than 96%. The 96% critical value was chosen so that the overall 1-sided Type I error was less than 10%; Test type: Non-Inferiority — Estimated by Bayesian beta-binomial model using non-informative uniform prior, ie, Beta (1,1), within individual induction arms. Posterior distribution of retention rate difference between arms was used to calculate posterior probability of NI of RI to SoC induction using a 10% NI margin or favorable trend of RI over SoC induction; Bayesian beta-binomial model = 11.82, 95% CI 2-sided [4.34 to 19.03] — Posterior probability of RI NI to SoC, ie, (RI - SoC)>10%=100.00%
Statistical Analysis 2: Comparison: Induction Phase: Rapid Induction vs Induction Phase: Standard of Care Induction; If the non-inferiority of rapid induction (RI) to standard of care (SoC) induction was declared, the posterior possibility of retention rate difference (RI - SoC) greater than 0 was estimated to evaluate the superiority of RI over SoC induction; Test type: Superiority — The posterior possibility of retention rate difference (RI - SoC) greater than 0 was estimated to evaluate the superiority of RI over SoC induction; Bayesian beta-binomial model = 11.82, 95% CI 2-sided [4.34 to 19.03] — Posterior probability that RI treatment is superior to SoC treatment=99.90%

3. Secondary Outcome: Maintenance Phase: Percentage of Days Opioids Were Used Over Weeks 10 to 38
Description: Participants' percentage of days opioids were used out of days assessed over Weeks 10 to 38 (inclusive), based on the TLFB for the prior week.
Time Frame: Weeks 10 to 38
Population: Full Analysis Set (FAS): Participants who met all inclusion/exclusion criteria, were randomised, and received at least 1 maintenance RBP-6000 injection post DB Randomisation. Participants were analysed according to the randomised treatment arm. This population served as the primary analysis population for efficacy analyses.
Measure: Mean (Standard Deviation); unit: Participants' Percentage of Days
Arm/Group | Maintenance Phase: Extended-release Buprenorphine 100 mg | Maintenance Phase: Extended-release Buprenorphine 300 mg
Number analyzed (Participants) | 218 | 216
Participants' Percentage of Days | 17.7 (27.80) | 15.9 (26.13)
Statistical Analysis 1: Comparison: Maintenance Phase: Extended-release Buprenorphine 100 mg vs Maintenance Phase: Extended-release Buprenorphine 300 mg; Test type: Superiority — A Wilcoxon rank sum test (Van Elteren 1960) stratified for randomisation factors was performed to compare the difference between the 2 treatment arms. The test result P-value was used inferentially, if the primary endpoint test was statistically significant; p = 0.8836, Wilcoxon rank sum (Van Elteren); Wilcoxon rank sum test stratified by DB randomisation factor (Van Elteren, 1960); Mean Difference (Net) = -1.73, 95% CI 2-sided [-6.83 to 3.36] — Van Elteren Test Z-Score for Difference Between Arms (300 mg - 100 mg)=-0.1464

4. Secondary Outcome: Maintenance Phase: Percentage of Responders for Weekly Opioid Use Over Weeks 10 to 38
Description: A responder for weekly opioid use is defined as a participant whose percentage of visits with opioid abstinence is greater than or equal to 80% over Weeks 10 to 38 inclusive.
  Opioid abstinence is defined as a negative urine drug screen (UDS) result and negative responses to the TimeLine Follow Back (TLFB) interview for opioid use. The TLFB asks participants to retrospectively estimate their daily drug use for each of the past 7 days prior to the visit. Opioid use will be assessed at 15 visits between Weeks 10 and 38.
Time Frame: Weeks 10 to 38
Population: Full Analysis Set (FAS): Participants who met all inclusion/exclusion criteria, were randomized, and received at least 1 maintenance RBP-6000 injection post DB Randomization. Participants were analyzed according to the randomized treatment arm. This population served as the primary analysis population for efficacy analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Phase: Extended-release Buprenorphine 100 mg | Maintenance Phase: Extended-release Buprenorphine 300 mg
Number analyzed (Participants) | 218 | 216
Participants | 42 | 45
Statistical Analysis 1: Comparison: Maintenance Phase: Extended-release Buprenorphine 100 mg vs Maintenance Phase: Extended-release Buprenorphine 300 mg; Opioid abstinence between Weeks 10 to 38 (inclusive) was derived as the participant's number of visits with negative assessments (defined as negative UDS and TLFB for opioid use) divided by 15. Under this derivation, any missed or skipped visits were counted as positive, in accordance with the composite Intercurrent Events Strategy. The opioid use derivation at a specific visit was the same as that used for the primary efficacy endpoint; Test type: Other; p = 0.6111, Cochran-Mantel-Haenszel; CMH weighted treatment difference and p-value based on the CMH randomization stratified analysis using the Sato (1989) variance equation; CMH Difference = 1.26, 95% CI 2-sided [-3.61 to 6.13] — CMH weighted treatment difference and p-value based on the CMH randomization stratified analysis using the Sato (1989) variance equation

5. Secondary Outcome: Maintenance Phase: Percentage of Visits With Opioid Abstinence Over Weeks 10 to 38
Description: Opioid abstinence is defined as negative urine drug screen results and negative responses to the TimeLine Follow Back (TLFB) interview for opioids.
  The TLFB asks participants to retrospectively estimate their daily drug use for each of the past 7 days prior to the visit.
Time Frame: Weeks 10 to 38
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Participants' Percentage of Visits
Arm/Group | Maintenance Phase: Extended-release Buprenorphine 100 mg | Maintenance Phase: Extended-release Buprenorphine 300 mg
Number analyzed (Participants) | 218 | 216
Participants' Percentage of Visits | 31.1 (37.18) | 32.1 (36.94)
Statistical Analysis 1: Comparison: Maintenance Phase: Extended-release Buprenorphine 100 mg vs Maintenance Phase: Extended-release Buprenorphine 300 mg; Opioid abstinence between Weeks 10 to 38 (inclusive) was derived as his/her number of visits with negative assessments (defined as negative UDS and TLFB for opioid use) divided by 15. Under this derivation, any missed or skipped visits were counted as positive, in accordance with the composite intercurrent event strategy; Test type: Other; Mean Difference (Net) = 1.00, 95% CI 2-sided [-6.00 to 7.99]

6. Secondary Outcome: Maintenance Phase: Percentage of Responders for Weekly Opioid Use Over Weeks 30 to 38
Description: A responder for weekly opioid use is defined as a participant whose percentage of visits with opioid abstinence is greater than or equal to 80% for the last 5 visits planned for urine drug screen (UDS) and TimeLine Follow Back (TLFB) over Weeks 30 to 38 (inclusive).
  Opioid abstinence is defined as a negative UDS result and negative responses to the TLFB interview for opioid use. The TLFB asks participants to retrospectively estimate their daily drug use for each of the past 7 days prior to the visit.
Time Frame: Week 30 to 38
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Phase: Extended-release Buprenorphine 100 mg | Maintenance Phase: Extended-release Buprenorphine 300 mg
Number analyzed (Participants) | 218 | 216
Participants | 50 | 56
Statistical Analysis 1: Comparison: Maintenance Phase: Extended-release Buprenorphine 100 mg vs Maintenance Phase: Extended-release Buprenorphine 300 mg; Test type: Other; This endpoint was summarized similar to the analysis for #4 above. The opioid abstinence percentage for an individual participant was derived as his/her number of visits with negative assessments divided by 5; CMH Difference = 2.73, 95% CI 2-sided [-4.98 to 10.43] — CMH weighted treatment difference based on the CMH randomization stratified analysis using the Sato (1989) variance equation

7. Secondary Outcome: Maintenance Phase: Percentage of Responders for Daily Opioid Use
Description: A responder for daily opioid use is defined as a participant with 20% or less days of opioid use, based on the TimeLine Follow Backs (TLFBs) collected at the last 5 observed visits post randomization. The TLFB asks participants to retrospectively estimate their daily drug use for each of the past 7 days prior to the visit.
Time Frame: Week 30 to 38
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Phase: Extended-release Buprenorphine 100 mg | Maintenance Phase: Extended-release Buprenorphine 300 mg
Number analyzed (Participants) | 218 | 216
Participants | 166 | 165
Statistical Analysis 1: Comparison: Maintenance Phase: Extended-release Buprenorphine 100 mg vs Maintenance Phase: Extended-release Buprenorphine 300 mg; Test type: Other; CMH Difference = 0.15, 95% CI 2-sided [-7.49 to 7.78] — [estimate comment as in outcome 6, analysis 1]

8. Secondary Outcome: Maintenance Phase: Percentage of Visits With Opioid Abstinence Overall
Description: Opioid abstinence is defined as negative urine drug screen results and negative responses to the TimeLine Follow Back (TLFB) interview for opioids at all assessments between Weeks 2 and 38. The TLFB asks participants to retrospectively estimate their daily drug use for each of the past 7 days prior to the visit.
Time Frame: Week 2 to 38
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Participants' Percentage of Visits
Arm/Group | Maintenance Phase: Extended-release Buprenorphine 100 mg | Maintenance Phase: Extended-release Buprenorphine 300 mg
Number analyzed (Participants) | 218 | 216
Participants' Percentage of Visits | 30.5 (33.24) | 32.0 (33.46)
Statistical Analysis 1: Comparison: Maintenance Phase: Extended-release Buprenorphine 100 mg vs Maintenance Phase: Extended-release Buprenorphine 300 mg; Test type: Other; Mean Difference (Net) = 1.49, 95% CI 2-sided [-4.80 to 7.78]

9. Secondary Outcome: Maintenance Phase: Percentage of Days Opioids Were Used Overall
Description: For each participant, the percentage of days opioids were used out of days assessed over Weeks 2 to 38 (inclusive), based on the TimeLine Follow Back (TLFB) for the prior week of each visit.
Time Frame: Week 2 to 38
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Participants' Percentage of Days
Arm/Group | Maintenance Phase: Extended-release Buprenorphine 100 mg | Maintenance Phase: Extended-release Buprenorphine 300 mg
Number analyzed (Participants) | 218 | 216
Participants' Percentage of Days | 18.3 (25.14) | 17.6 (25.04)
Statistical Analysis 1: Comparison: Maintenance Phase: Extended-release Buprenorphine 100 mg vs Maintenance Phase: Extended-release Buprenorphine 300 mg; Test type: Other; Mean Difference (Net) = -0.64, 95% CI 2-sided [-5.38 to 4.09]

10. Secondary Outcome: Maintenance Phase: Percentage of Days Opioids Were Used Via the Injection Route
Description: For participants who use opioids via the injection route for an average of 5 or more days per week in the last 4 weeks prior to Screening, the percentage of days opioids were used via the injection route out of days assessed based on the Timeline Follow Back (TLFB) interview for the prior week of each visit.
Time Frame: Weeks 10 to 38
Population: Full Analysis Set (FAS) Subpopulation: Participants who met all inclusion/exclusion criteria, were randomized, and received at least 1 maintenance RBP-6000 injection post DB Randomization; for this analysis, only participants who use opioids via the injection route for an average of ≥5 days per week in the last 4 weeks prior to Screening were included. Participants were analyzed according to the randomized treatment arm.
Measure: Mean (Standard Deviation); unit: Participants' Percentage of Days
Arm/Group | Maintenance Phase: Extended-release Buprenorphine 100 mg | Maintenance Phase: Extended-release Buprenorphine 300 mg
Number analyzed (Participants) | 65 | 61
Participants' Percentage of Days | 9.9 (23.79) | 8.5 (19.01)
Statistical Analysis 1: Comparison: Maintenance Phase: Extended-release Buprenorphine 100 mg vs Maintenance Phase: Extended-release Buprenorphine 300 mg; Test type: Other; Mean Difference (Net) = -1.37, 95% CI 2-sided [-9.00 to 6.25]

11. Secondary Outcome: Maintenance Phase: Average Number of Times Opioids Were Used Per Week by Visit
Description: The average number of times opioids were used per week for a given visit based on the TimeLine Follow Back (TLFB) for the prior week collected at that visit.
Time Frame: Baseline to Week 38
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Ave Num of Times Opioids Were Used/Week
Arm/Group | Maintenance Phase: Extended-release Buprenorphine 100 mg | Maintenance Phase: Extended-release Buprenorphine 300 mg
Number analyzed (Participants) | 218 | 216
Ave Num of Times Opioids Were Used/Week
  Screening | 41.4 (32.08) | 44.9 (40.89)
  Week 1 Day 1: number analyzed (Participants) | 218 | 213
  Week 1 Day 1 | 26.3 (25.52) | 23.7 (26.90)
  Week 2: number analyzed (Participants) | 218 | 215
  Week 2 | 3.9 (9.58) | 4.6 (11.31)
  Week 3: number analyzed (Participants) | 210 | 210
  Week 3 | 2.4 (5.57) | 2.8 (6.66)
  Week 6: number analyzed (Participants) | 217 | 215
  Week 6 | 3.2 (7.69) | 4.0 (8.46)
  Week 10: number analyzed (Participants) | 202 | 201
  Week 10 | 3.2 (9.72) | 2.8 (5.51)
  Week 20: number analyzed (Participants) | 168 | 160
  Week 20 | 3.6 (11.35) | 2.3 (5.34)
  Week 34: number analyzed (Participants) | 140 | 140
  Week 34 | 3.1 (9.21) | 3.2 (10.36)
  Week 38/End of Treatment: number analyzed (Participants) | 134 | 125
  Week 38/End of Treatment | 2.8 (8.94) | 2.4 (8.71)

12. Secondary Outcome: Maintenance Phase: Change From Baseline in Number of Times Opioids Were Used Per Week
Description: The change in participants' number of times opioids were used per week from randomization baseline to each visit based on the 7 daily TimeLine Follow Back (TLFB) for the prior week collected at that visit.
Time Frame: Baseline to Week 38
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: % Change from Screening
Arm/Group | Maintenance Phase: Extended-release Buprenorphine 100 mg | Maintenance Phase: Extended-release Buprenorphine 300 mg
Number analyzed (Participants) | 218 | 216
% Change from Screening
  Week 1 Day 1: number analyzed (Participants) | 190 | 189
  Week 1 Day 1 | -30.7 (63.88) | -40.4 (52.63)
  Week 2: number analyzed (Participants) | 209 | 209
  Week 2 | -88.4 (25.81) | -88.6 (26.09)
  Week 3: number analyzed (Participants) | 162 | 163
  Week 3 | -94.3 (13.18) | -92.5 (19.00)
  Week 6: number analyzed (Participants) | 166 | 173
  Week 6 | -91.3 (18.91) | -90.6 (18.63)
  Week 10: number analyzed (Participants) | 161 | 158
  Week 10 | -92.9 (18.67) | -91.1 (17.12)
  Week 20: number analyzed (Participants) | 165 | 159
  Week 20 | -92.4 (17.03) | -93.2 (15.46)
  Week 34: number analyzed (Participants) | 137 | 139
  Week 34 | -93.5 (17.59) | -88.9 (46.94)
  Week 38/End of Treatment: number analyzed (Participants) | 132 | 124
  Week 38/End of Treatment | -93.6 (16.51) | -92.5 (24.89)

13. Secondary Outcome: Maintenance Phase: Percentage of Participants Who Were Opioid Abstinent by Visit
Description: Opioid abstinence is defined as negative urine drug screen results and negative responses to the TimeLine Follow Back (TLFB) interview for opioids.
Time Frame: Baseline to Week 38
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Phase: Extended-release Buprenorphine 100 mg | Maintenance Phase: Extended-release Buprenorphine 300 mg
Number analyzed (Participants) | 218 | 216
Participants
  Screening | 0 | 0
  Week 1 Day 1: number analyzed (Participants) | 218 | 215
  Week 1 Day 1 | 11 | 14
  Week 2 | 40 | 51
  Week 3: number analyzed (Participants) | 212 | 210
  Week 3 | 56 | 66
  Week 6 | 67 | 65
  Week 10: number analyzed (Participants) | 202 | 203
  Week 10 | 73 | 77
  Week 20: number analyzed (Participants) | 169 | 162
  Week 20 | 67 | 65
  Week 34: number analyzed (Participants) | 140 | 140
  Week 34 | 57 | 68
  Week 38/End of Treatment: number analyzed (Participants) | 134 | 128
  Week 38/End of Treatment | 63 | 64

14. Secondary Outcome: Maintenance Phase: Average Number of Days Opioids Were Used Per Week by Visit
Description: The average number of days opioids were used per week out of days assessed, based on the TimeLine Follow Back (TLFB) for the prior week of each visit.
Time Frame: Baseline to Week 38
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Average Number of Days
Arm/Group | Maintenance Phase: Extended-release Buprenorphine 100 mg | Maintenance Phase: Extended-release Buprenorphine 300 mg
Number analyzed (Participants) | 218 | 216
Average Number of Days
  Screening | 6.7 (0.97) | 6.9 (0.57)
  Week 1 Day 1: number analyzed (Participants) | 218 | 213
  Week 1 Day 1 | 5.1 (2.52) | 4.9 (2.60)
  Week 2: number analyzed (Participants) | 218 | 215
  Week 2 | 1.7 (2.18) | 1.7 (2.15)
  Week 3: number analyzed (Participants) | 210 | 210
  Week 3 | 1.3 (1.94) | 1.2 (1.94)
  Week 6: number analyzed (Participants) | 217 | 215
  Week 6 | 1.6 (2.18) | 1.4 (2.13)
  Week 10: number analyzed (Participants) | 202 | 201
  Week 10 | 1.3 (2.07) | 1.3 (2.14)
  Week 20: number analyzed (Participants) | 168 | 160
  Week 20 | 1.3 (2.21) | 1.0 (1.85)
  Week 34: number analyzed (Participants) | 140 | 140
  Week 34 | 1.2 (2.21) | 0.9 (1.98)
  Week 38/End of Treatment: number analyzed (Participants) | 134 | 125
  Week 38/End of Treatment | 1.2 (2.24) | 0.9 (2.07)

15. Secondary Outcome: Maintenance Phase: Time From DB Randomization to Last Observed Study Visit (Treatment Retention)
Description: Treatment retention is defined as the number of days that participants remained in the treatment from randomization in the Maintenance Phase of the study until the date of the last observed study visit.
  The treatment retention since DB randomization is estimated using Kaplan-Meier method. The event is prematurely discontinuing the study prior to Week 38/EOT Visit.
Time Frame: Up to 288 days after randomization (accounting for out-of-window visits)
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Maintenance Phase: Extended-release Buprenorphine 100 mg | Maintenance Phase: Extended-release Buprenorphine 300 mg
Number analyzed (Participants) | 218 | 216
Days | 266 [241 to NA] — NA Explanation: the 95% upper confidence limit for the median is not estimable by the Kaplan-Meier method because the curve representing the upper confidence intervals for the survivor function lies above 0.50. | 260 [113 to NA] — NA Explanation: the 95% upper confidence limit for the median is not estimable by the Kaplan-Meier method because the curve representing the upper confidence intervals for the survivor function lies above 0.50.

16. Secondary Outcome: Maintenance Phase: Percentage of Participants Who Complete the Last Scheduled Injection
Description: The proportion of randomized participants who completed the last scheduled injection of RBP-6000 at Week 34 were summarized using observed data. Missing data were not applicable for this endpoint.
Time Frame: Week 34
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Phase: Extended-release Buprenorphine 100 mg | Maintenance Phase: Extended-release Buprenorphine 300 mg
Number analyzed (Participants) | 218 | 216
Participants | 138 | 140
Statistical Analysis 1: Comparison: Maintenance Phase: Extended-release Buprenorphine 100 mg vs Maintenance Phase: Extended-release Buprenorphine 300 mg; Test type: Other; CMH Difference = 1.54, 95% CI 2-sided [-7.56 to 10.65] — CMH weighted treatment difference based on the CMH randomisation stratified analysis using the Sato (1989) variance equation

17. Secondary Outcome: Induction Phase: Percentage of Participants Retained at 5 Weeks
Description: Percentage of participants retained at 5 weeks after the first dose of TM buprenorphine was estimated using the Kaplan-Meier product limit method.
Time Frame: 35 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Induction Phase: Rapid Induction | Induction Phase: Standard of Care Induction
Number analyzed (Participants) | 470 | 253
Percentage of participants | 60.2 [55.6 to 64.5] | 53.4 [47.0 to 59.3]
Statistical Analysis 1: Comparison: Induction Phase: Rapid Induction vs Induction Phase: Standard of Care Induction; Test type: Other; Cox Proportional Hazard = 0.82, 95% CI 2-sided [0.65 to 1.03] — Estimated using a Cox proportional hazard model, with treatment arm as a single covariate, stratified by the randomisation strata. Note that the estimation is impacted by last observed visit for the OLTP (including out-of-window visits)

18. Secondary Outcome: Induction Phase: Number of Participants With Adverse Events up to Injection 2
Description: These endpoints encompassed all induction attempts and therefore utilized the first dose of transmucosal buprenorphine (TM BUP) for derivations. A treatment-emergent adverse event (TEAE) was defined as an AE having an onset date/time after administration of the first TM BUP dose and before the date/time of Injection 3. TEAEs up to RBP-6000 Injection 2 were TEAEs with a start date/time on or after the first dose of TM BUP and before the date/time of Injection 2.
Time Frame: Up to approximately 2 weeks
Population: Substudy Full Analysis Set (SFAS): All participants randomized to open-label substudy treatment, received the first dose of TM BUP, and did not demonstrate idiosyncratic response to the first dose of TM BUP (ie, allergic / hypersensitivity reaction). Participants were analyzed corresponding to the induction arm they received ("as treated", ie, actual arm).
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Phase: Rapid Induction | Induction Phase: Standard of Care Induction
Number analyzed (Participants) | 474 | 255
Participants | 202 | 93

19. Secondary Outcome: Induction Phase: Number of Participants With Adverse Events Between Injections 2 and 3
Description: These endpoints encompassed all induction attempts and therefore utilized the first dose of transmucosal buprenorphine (TM BUP) for derivations. A treatment-emergent adverse event (TEAE) was defined as an AE having an onset date/time after administration of the first TM BUP dose and before the date/time of Injection 3. TEAEs between RBP-6000 Injections 2 and 3 were TEAEs with a start date/time on or after Injection 2 and before the date/time of Injection 3.
Time Frame: Approximately 4 weeks
Population: Substudy Full Analysis Set (SFAS): All participants randomized to open-label substudy treatment, received the first dose of TM BUP, and did not demonstrate idiosyncratic response to the first dose of TM BUP (ie, allergic / hypersensitivity reaction). Participants were analyzed corresponding to the induction arm they received ("as treated", ie, actual arm). For this analysis, only SFAS participants who received Injection 2 were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Phase: Rapid Induction | Induction Phase: Standard of Care Induction
Number analyzed (Participants) | 314 | 138
Participants | 86 | 29

ADVERSE EVENTS:
Time Frame: Approximately 38 weeks
Description: Investigator or designee was responsible for identifying, documenting, and reporting events that met the AE definition. The Open-label Induction Substudy (OLIS) and main study were reported separately (ie, Induction [Rapid Induction vs Standard of Care Induction] and Maintenance [100 mg vs 300 mg]).
  Induction Phase (OLIS) used MedDRA 26.1 and Double-blind Treatment Phase (Injection 3 through the end of the study) used MedDRA 27.0.
  SAEs were not subtracted from other AEs for "Other" AE table.
Arm/Group | Induction Phase: Rapid Induction | Induction Phase: Standard of Care Induction | Maintenance Phase: Extended-release Buprenorphine 100 mg | Maintenance Phase: Extended-release Buprenorphine 300 mg
All-Cause Mortality (participants affected / at risk) | 1/474 | 0/255 | 0/218 | 1/217
Serious Adverse Events (participants affected / at risk) | 7/474 | 1/255 | 11/218 | 11/217
Other Adverse Events (participants affected / at risk) | 135/474 | 58/255 | 11/218 | 30/217
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Phase: Rapid Induction (N=474) | Induction Phase: Standard of Care Induction (N=255) | Maintenance Phase: Extended-release Buprenorphine 100 mg (N=218) | Maintenance Phase: Extended-release Buprenorphine 300 mg (N=217)
Sedation (Nervous system disorders) | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Drug withdrawal syndrome (General disorders) | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1
Brain abscess (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Intentional self-injury (Psychiatric disorders) | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Transient ischemic attack (Nervous system disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Phase: Rapid Induction (N=474) | Induction Phase: Standard of Care Induction (N=255) | Maintenance Phase: Extended-release Buprenorphine 100 mg (N=218) | Maintenance Phase: Extended-release Buprenorphine 300 mg (N=217)
Nausea (Gastrointestinal disorders) | 65 | 31 | 0 | 0
Vomiting (Gastrointestinal disorders) | 32 | 15 | 0 | 0
Anxiety (Psychiatric disorders) | 50 | 21 | 0 | 0
Restlessness (Psychiatric disorders) | 33 | 14 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 26 | 11 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 6 | 11
Vomiting (Gastrointestinal disorders) | 0 | 0 | 4 | 13
Injection site pain (General disorders) | 0 | 0 | 3 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator will not disseminate, present or publish any of the study data without the prior written approval from Indivior to do so.

DOCUMENTS (3):
  • Study Protocol (2022-04-07): https://cdn.clinicaltrials.gov/large-docs/29/NCT04995029/Prot_000.pdf
  • Statistical Analysis Plan: Main Study - Double-blind Maintenance Phase (2024-08-22): https://cdn.clinicaltrials.gov/large-docs/29/NCT04995029/SAP_001.pdf
  • Statistical Analysis Plan: Open-label Induction Study (2023-08-25): https://cdn.clinicaltrials.gov/large-docs/29/NCT04995029/SAP_002.pdf